CLINICAL TRIAL: NCT03847948
Title: Evaluation of Biological Factors Associated With Subclinical Valvular Thrombosis in pAtients With Severe aoRtic Stenosis Undergoing TAVI: START Trial
Brief Title: Biological Factors Associated With Subclinical Valvular Thrombosis
Acronym: START
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Pilar Jimenez Quevedo, MD, PhD, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: PI17/01685
Record Dates: First submitted 2019-02-03; First posted 2019-02-20 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, multicentric cohort study including 166 patients with symptomatic aortic stenosis treated with transcatheter aortic valve implantation (TAVI).

- The main objective is to determine whether the high residual platelet reactivity rates in patients undergoing TAVI is associated with the occurrence of clinical and / or subclinical prosthetic valve thrombosis measured by echocardiography and multi-slice computerized tomography

DETAILED DESCRIPTION:
For the purpose of the study, platelet reactivity will be measured with the commercial kit PLT VASP/P2Y12 at baseline, 1day and 3 months postprocedure.

Secondary objectives include: -Determine the variability of platelet aggregation measured at baseline before the procedure, 1-day post-procedure and at 3-6 and 1 year follow-up.

* To determine whether the pro-thrombotic inflammatory response measured by the CD14 + and CD16 + quantification observed after TAVI is associated with the appearance of prosthetic thrombosis.
* To evaluate the Correlation of Von Willebrand factor levels and distribution of Von Willebrand multimers with the appearance of prosthetic thrombosis at baseline before the procedure, 1-day post-procedure and at 3, 6 months follow-up and 1 year.
* To determine whether the residual platelet reactivity rates in patients undergoing TAVI are associated with the occurrence of clinical events, at baseline before the procedure, 1-day post-procedure and at 3,6 months follow-up and 1 year
* To evaluate the clinical factors associated with the appearance of early prosthetic thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe symptomatic aortic stenosis who it was accepted to be treated with TAVI by a multidisciplinary team "Heat Team".
* TAVI was successfully implanted (according to Valve Academic Research Consortium II criteria) and are under treatment with double antiplatelet therapy.
* Signed informed consent to participate in this study.

Exclusion Criteria:

* Age under 18 years and pregnant or of childbearing age.
* Acute Recent stroke recent <14 days before TAVI.
* The patients with proven allergy to aspirin, clopidogrel
* Patients that after TAVI cannot undergo a double antiplatelet regimen for 6 months due to a new post-TAVI medical indication or are anticoagulated.
* Knowledge of pregnancy or lactation Thrombocytopenia (<50,000 platelets U / L) well documented and clinically relevant.
* The patients with documented moderate or severe hepatic insufficiency
* Severe chronic renal insufficiency with creatinine clearance <30 ml / min.
* The patients who can not attend the follow-up visits scheduled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic aortic stenosis treated with TAVI
Sampling Method: Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
The association between high residual platelet reactivity rates in patients undergoing TAVI with the occurrence of clinical and / or subclinical prosthetic valve thrombosis | at 3 months
  platelet reactivity will be measured with the commercial kit platelet Vasodilator Stimulated Phosphoprotein (VASP)/P2Y12 and subclinical valve thrombosis by transthoracic echocardiography and multi-slice computerized tomography

SECONDARY OUTCOMES:
To measure the variability of platelet aggregation | at baseline, 1 day post-procedure and at 3-6 months and 1 year follow-up.
  platelet aggregation
To quantify the pro-thrombotic inflammatory response | at baseline, 1 day post-procedure and at 3, 6 months and 1 year follow-up.
  measured by serum levels of (cluster of differentiation 14) CD14 + and (cluster of differentiation 16) CD16 +
To correlate of Von Willebrand factor levels and distribution of Von Willebrand factor multimers with the appearance of prosthetic thrombosis | at baseline, 1 day post-procedure and at 3, 6 months and 1 year follow-up.
  Serum Von Willebrand factor levels and distribution of Von Willebrand factor multimers with the appearance of prosthetic thrombosis assessed by transthoracic echocardiography or multi-slice computerized tomography
To correlate residual platelet reactivity with clinical events | at baseline, 1 day post-procedure and at 3, 6 months and 1 year follow-up.
  platelet aggregation
To evaluate clinical factors associated with the appearance of early prosthetic thrombosis. | multi slice computerized tomography at 3 month and clinical up to 1 year.
  to perform Multislice computerized tomography and clinical follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clinic, Barcelona
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No